CLINICAL TRIAL: NCT04698278
Title: Post-Approval Study of the Panoptix Trifocal Lens in Patients Who Have Had Post Refractive Myopic Laser Vision Correction Surgery
Brief Title: Panoptix Trifocal Lens in Post Refractive Myopic Laser Vision Correction Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parkhurst NuVision Clinical Research LLC (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Brett Mueller, Principal Investigator, Parkhurst NuVision Clinical Research LLC
Other Study IDs: TFL210
Record Dates: First submitted 2020-12-02; First posted 2021-01-06 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cataract; Refractive Errors
MeSH Terms: conditions — Cataract; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Surgical Treatment Group: This is a prospective, single center, bilateral, non-randomized, open-label, observational clinical study. All patients will have had prior myopic Lasik and will receive a PanOptix Trifocal IOL in both eyes at the time of cataract surgery. These patients will then be followed for up to 6-months to assess their refractive predictability, quality of vision, spectacle independence, and overall patient satisfaction.
  Interventions: Device: PanOptix Trifocal Intraocular Lens

INTERVENTIONS:
Device: PanOptix Trifocal Intraocular Lens — This is a FDA approved trifocal lens that will be placed in patients who have had previous myopic LASIK or PRK.

SUMMARY:
The two main objectives of this study are to demonstrate safety and effectiveness of implanting the PanOptix Trifocal IOL in patients who have had previous myopic Lasik. The primary objectives to demonstrate clinical safety will be the quality of vision questionnaire (QUVID) which will demonstrate the patient's perception of halos, glares, and starbursts before and after the implantation of the trifocal IOL.

The primary objective to demonstrate clinical effectiveness will be done by measuring visual outcomes at distance, intermediate, and near. In addition, the patients will also fill out the spectacle independence questionnaire (IOLSAT Questionnaire) to determine their level of glasses independence postoperatively. In addition, at the conclusion of the study the patient will also fill out a patient satisfaction survey.

DETAILED DESCRIPTION:
Clinical Hypothesis:

The rate of bothersome visual symptom items (defined as a very or extremely bothersome visual symptom that impacts daily living under overall condition) for the patients who are post-refractive who receive a PanOptix Trifocal IOL at the time of cataract surgery will be assessed. The bothersome visual symptom items of interest are halos, glare, and starbursts. Patients will also be assessed on level of glasses independence with an assessment of both corrected and uncorrected distance, intermediate, and near vision. Lastly patient satisfaction score will also be determined.

OVERALL STUDY DESIGN This is a prospective, single center, bilateral, non-randomized, open-label, observational clinical study. All patients will have had prior myopic Lasik and will receive a PanOptix Trifocal IOL in both eyes at the time of cataract surgery. These patients will then be followed for up to 6-months to assess their refractive predictability, quality of vision, spectacle independence, and overall patient satisfaction.

Duration:

6 months; however, any subject that undergoes a lens repositioning procedure due to IOL misalignment, or reports "very" or "extreme" overall bother that impacts daily living for any of the 3 defined bothersome visual symptoms (halos, glare, or starbursts) at 6 months, will be followed through 1 year postoperatively.

Administration:

Surgeons will perform routine small-incision, femtosecond laser assisted, cataract surgery and use the Alcon-recommended implantation systems for lens implantation. Refractive target outcomes will be emmetropia for both eyes.

Visit Schedule:

Subjects will be bilaterally implanted; the second eye is to be implanted within approximately one month after the first-eye surgery.

All subjects will undergo a minimum of 10 visits:

1. Preoperative for both eyes
2. Surgical Procedure for each individual eye
3. 1-day and 1-week visits for each eye
4. 1-month, 3-month, and 6-month visits for both eyes together
5. In addition, a 1-year postoperative visit will be required for subjects who undergo a lens repositioning procedure due to IOL misalignment at any time during the study, and for subjects who report "very" or "extreme" overall bother that impacts daily living for any of the 3 defined bothersome visual symptoms (halos, glare, or starbursts) at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 22 years of age or older at the time of surgery, diagnosed with bilateral cataracts with planned cataract removal by phacoemulsification with a clear cornea incision
2. Previous myopic Lasik with a well centered optical zone, corneal higher-order aberrations less than 0.6 um for a 4 mm pupil (measured by iTrace), and a minimum keratometric reading of 35.0 D.
3. Able to comprehend and willing to sign informed consent and complete all required postoperative follow-up procedures
4. Best Corrected Distance Visual Acuity (BCDVA) projected to be 0.2 logMAR (Minimum Angle of Resolution) or better
5. Calculated lens power within the available range
6. Preoperative keratometric astigmatism at or less than 2.5 D in both operative eyes
7. Clear intraocular media other than cataract in both eyes

Exclusion Criteria:

1. Clinically significant corneal abnormalities including corneal dystrophy, irregularity, inflammation or edema.
2. Previous intraocular surgery other than myopic Lasik
3. History of or current retinal conditions or predisposition to retinal conditions
4. Amblyopia
5. Rubella, congenital, traumatic, or complicated cataracts
6. History of or current anterior or posterior segment inflammation of any etiology
7. Iris neovascularization
8. Glaucoma (uncontrolled or controlled with medication)
9. Optic nerve atrophy
10. Subjects with diagnosed degenerative eye disorders
11. Pregnancy or lactation
12. Any disease or pathology, other than cataract, that is expected to reduce the potential postoperative BCDVA to a level worse than 0.30 logMAR.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bilateral cataracts in individuals who have had prior myopic laser assisted in situ keratomileusis or photorefractive keratectomy. Topography ablation patterns need to be well centered, and the corneal higher order aberration number needs to be less than 0.6 um for a 4 mm pupillary diameter on the itrace. PanOptix IOL power will be selected by utilizing the American Society of Cataract and Refractive Surgery online post refractive calculator: https://iolcalc.ascrs.org/. In addition, this IOL power calculation will be confirmed with Alcon's intraoperative ORA aberrometer.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Quality of vision questionnaire (QUVID) | 3 months post surgery
  Will assess patient complaints of glares, halos and starbursts after implantation of the trifocal PanOptix lens. Each of these three symptoms will be assessed on how often they occur, severity of each symptom, and how bothersome they are for the patient. The patient will rank the how often they occur as never, rarely, sometimes, most of the time, and always. The patient will rank severity of their worst experience as: none, a little, mild, moderate, and severe. And the patient will rank how bothered they are by each of these symptoms as: not bothered at all, bothered a little bit, bothered somewhat, bothered quite a bit, or bothered very much.
Quality of vision questionnaire (QUVID) | 6 months post surgery
  Will assess patient complaints of glares, halos and starbursts after implantation of the trifocal PanOptix lens. Each of these three symptoms will be assessed on how often they occur, severity of each symptom, and how bothersome they are for the patient. The patient will rank the how often they occur as never, rarely, sometimes, most of the time, and always. The patient will rank severity of their worst experience as: none, a little, mild, moderate, and severe. And the patient will rank how bothered they are by each of these symptoms as: not bothered at all, bothered a little bit, bothered somewhat, bothered quite a bit, or bothered very much.
Patient Vision Satisfaction Survey | 3 months post surgery
  Will look at the level of patient satisfaction with their overall visual quality. Patient will be asked to grade their visual satisfaction as being very satisfied, satisfied, neither satisfied nor dissatisfied, or dissatisfied.
Patient Vision Satisfaction Survey | 6 months post surgery
  Will look at the level of patient satisfaction with their overall visual quality. Patient will be asked to grade their visual satisfaction as being very satisfied, satisfied, neither satisfied nor dissatisfied, or dissatisfied.
Spectacle Independence Questionnaire (IOLSAT Questionnaire) | 3 months post surgery
  Will look at the level of spectacle independence in patients who receive the trifocal PanOptix IOL for their cataracts. Patients will be asked how often they need to wear glasses for near, intermediate, and distant activities in both dim and bright lighting conditions. These will be graded as rarely, sometimes, most of the time, and all the time. Patients will also be asked to characterize their overall visual quality without glasses at near, intermediate, and distant activities in dim and bright lighting conditions. Patients will rank these as: very poor, poor, fair, good, or very good.
Spectacle Independence Questionnaire (IOLSAT Questionnaire) | 6 months post surgery
  Will look at the level of spectacle independence in patients who receive the trifocal PanOptix IOL for their cataracts. Patients will be asked how often they need to wear glasses for near, intermediate, and distant activities in both dim and bright lighting conditions. These will be graded as rarely, sometimes, most of the time, and all the time. Patients will also be asked to characterize their overall visual quality without glasses at near, intermediate, and distant activities in dim and bright lighting conditions. Patients will rank these as: very poor, poor, fair, good, or very good.
Mean photopic monocular and binocular best corrected and uncorrected visual acuity at distance (6 meters), intermediate (60 cm), and near (40 cm). | 3 months post surgery
  Will assess vision at these 3 focal points
Mean photopic monocular and binocular best corrected and uncorrected visual acuity at distance (6 meters), intermediate (60 cm), and near (40 cm). | 6 months post surgery
  Will assess vision at these 3 focal points

CONTACTS AND LOCATIONS:
Locations (1):
- Parkhurst NuVision, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to present this data at research meetings and in research journals pertinent to ophthalmology.